CLINICAL TRIAL: NCT06924450
Title: Effect of Modified Mesh on Surgical Success in Transobturator Tape Surgery
Acronym: MOTOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izzet Celegen (Other)
Responsible Party: Sponsor-Investigator, Izzet Celegen, Assistant professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YB-MESH-2025-VAN001; EK-090523 (Other: Van Regional Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-02-24; First posted 2025-04-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stress Urinary Incontinence; Female Urinary Incontinence; Pelvic Floor Dysfunction
Keywords: Urinary Incontinence; Stress Urinary Incontinence (SUI); Female Pelvic Health; Transobturator Tape (TOT) Procedure; Pelvic Floor Surgery; Surgical Mesh; Randomized Controlled Trial; Urogynecology
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: This randomized, single-blind parallel-group study compares the surgical outcomes of two mesh widths (1.2 cm vs. 1.0 cm) used in transobturator tape (TOT) surgery for women with stress urinary incontinence (SUI).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor evaluating postoperative results is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.2 cm Mesh (Intervention Group) (Experimental): Participants in this group will undergo transobturator tape (TOT) surgery using a 1.2 cm monofilament polypropylene mesh.
  Interventions: Device: 1.2 cm Mesh TOT
- 1.0 cm Mesh (Control Group) (Active Comparator): Participants in this group will undergo transobturator tape (TOT) surgery using a 1.0 cm monofilament polypropylene mesh, which represents the standard procedure.
  Interventions: Device: 1.0 cm Mesh TOT

INTERVENTIONS:
Device: 1.2 cm Mesh TOT — Patients in this group will undergo transobturator tape (TOT) surgery using a 1.2 cm monofilament polypropylene mesh. The modified mesh width is being evaluated for its effect on surgical success, symptom improvement, and postoperative complications.
  Arms: 1.2 cm Mesh (Intervention Group)
Device: 1.0 cm Mesh TOT — Patients in this group will undergo transobturator tape (TOT) surgery using a 1.0 cm monofilament polypropylene mesh, which is the standard procedure. This group serves as a comparator to assess the impact of the modified mesh width.
  Arms: 1.0 cm Mesh (Control Group)

SUMMARY:
This study is a single-blind, randomized controlled trial evaluating whether changing the width of the surgical tape (mesh) used in transobturator tape (TOT) surgery improves treatment results in women with stress urinary incontinence (SUI). Two mesh widths are being compared: a 1.2 cm mesh (new method) and a 1.0 cm mesh (standard method). The main goal is to find out if the wider mesh leads to better urinary control and fewer complications. Participants will be followed for one year to measure cure rates, symptom improvement, and satisfaction.

DETAILED DESCRIPTION:
This is a prospective, single-blind, randomized controlled trial evaluating the effect of mesh width on surgical outcomes in transobturator tape (TOT) procedures for women with stress urinary incontinence (SUI). A total of 106 participants will be randomized using a computer-generated allocation into two groups receiving either a 1.2 cm mesh (intervention group) or a 1.0 cm mesh (standard procedure).

The procedures will be conducted by a single experienced surgeon using a monofilament polypropylene mesh to ensure standardization. Surgical technique, anesthesia protocols, and perioperative management will be identical in both groups.

Primary outcome is objective cure, defined as negative stress test at 6 months. Secondary outcomes include symptom improvement (ICIQ-SF), mesh-related complications (erosion, infection, retention), and patient satisfaction assessed via structured Likert survey.

Follow-up visits are scheduled at 1 week, 1 month, and 1 year. Postoperative assessments will be conducted by a blinded evaluator. The study aims to evaluate whether wider mesh width provides superior anatomical support and reduces complication rates in comparison to standard mesh.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Clinical diagnosis of stress urinary incontinence (SUI), confirmed by:
* Positive stress test (urine leakage on coughing with a comfortably full bladder)
* Q-tip test showing urethral hypermobility (>30 degrees)
* Inadequate response to conservative therapy (e.g., pelvic floor muscle training, behavioral therapy)
* Eligible for transobturator tape (TOT) surgery
* Body mass index (BMI) less than 35 kg/m²
* Able to provide informed consent and follow postoperative instructions

Exclusion Criteria:

* History of prior midurethral sling surgery
* Mixed urinary incontinence or urge-dominant symptoms
* Pelvic organ prolapse stage > II according to the POP-Q system
* Neurological disorders affecting bladder function (e.g., multiple sclerosis, spinal cord injury)
* Active urinary tract infection or recurrent UTI (defined as ≥3 infections within the past 12 months)
* Pregnant or planning to become pregnant within the next 12 months
* Severe comorbid conditions (e.g., uncontrolled diabetes mellitus, active malignancy, pelvic radiotherapy)
* Use of medications that significantly affect bladder function (e.g., anticholinergics, diuretics)
* Inability or unwillingness to attend follow-up visits or comply with postoperative care plan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Objective Cure Rate Based on Negative Stress Test | 6 months postoperatively
  Objective cure will be defined as the absence of urinary leakage during a standardized cough stress test with a comfortably full bladder. The test will be performed by a blinded assessor at 6 months postoperatively.

SECONDARY OUTCOMES:
Change in ICIQ-SF Score | 6 months postoperatively
  Change in total score on the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), measured before surgery and at 6 months postoperatively. The ICIQ-SF ranges from 0 to 21, with higher scores indicating worse symptom severity and greater impact on quality of life.
Incidence of Mesh-Related Complications | 6 months postoperatively
  Incidence of mesh-related complications including mesh erosion, bladder outlet obstruction, infection, and pain. Complications will be assessed by physical examination and patient-reported symptoms during follow-up visits.
Recurrence of Stress Urinary Incontinence | 6 months postoperatively
  Proportion of patients who present with recurrence of stress urinary incontinence, defined as a positive cough stress test or self-reported symptoms of urine leakage during physical activity.
  Time Frame: 6 months postoperatively
Patient Satisfaction Score | 6 months postoperatively
  Patient satisfaction will be measured using a structured questionnaire that includes a 5-point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied). Higher scores indicate greater satisfaction. Assessment will be conducted at the 6-month follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Regional Training and Research Hospital, Department of Obstetrics and Gynecology, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to confidentiality policies and institutional regulations. Summary-level results may be shared upon request.